CLINICAL TRIAL: NCT05751174
Title: Determination of Nerve Growth Factor (NGF) Expression in Pediatric Patients With Severe Burns: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Conti Giorgio, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3935
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Burns
Keywords: nerve growth factor; pediatric patient
MeSH Terms: conditions — Burns; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pediatric patients affected by severe burns — All patients admitted to the pediatric intensive care unit affected by severe burns involving more than 10% of the body surface will be enrolled.

SUMMARY:
The goal of this observational study is to determine the blood values of NGF in severely burned patients, to describe any changes over time and finally to correlate the expression of NGF to the severity of the burn.

The main question it aims to answer is:

- describe NGF values in severely burned pediatric patients and to evaluate their correlation with the severity of the burn and the extent of the burned skin surface by measuring the circulating levels of NGF in pediatric patients.

Participants will undergo blood sampling on days 2,7,14 and 30 after the traumatic event for the clinical follow-up envisaged by the internal protocol.

DETAILED DESCRIPTION:
Severe pediatric burns, characterized by an extension greater than 10% of the total body surface or by the involvement of particular districts such as the hands, face, airways or genitals, are characterized by multisystem involvement, which often requires intensive care support.

The epidermis begins to develop from the superficial ectoderm at the end of the fourth week of gestation when the neural tube separates from the overlying ectoderm. Consequently, the ectoderm gives rise to both the nervous system and the epithelium.

In particular, the NERVE GROWTH FACTOR (NGF) is a neurotrophic factor that plays a fundamental protective role in the development and survival of neurons.

In fetal skin, NGF is synthesized in both the epithelium and mesenchyme, but the highest amounts of NGF messenger ribonucleic acid are found in the epithelium. There are currently no studies investigating the expression of NGF in severe burns.

The common embryonic origin of the skin and the neurological system may hold the key to new research opportunities to understand the regenerative response and in particular the role of growth factors such as NGF in the skin repair mechanism in severe burns .

The hypothesis of the study is based on the possibility that skin burns may be related to an increased expression of circulating NGF in the blood. However, there are no data in literature on this issue and the behavior of NGF in patients affected by burns is not known, either in adult or pediatric patients.

Aim To describe NGF values in severely burned pediatric patients and to evaluate their correlation with the severity of the burn and the extent of the burned skin surface by measuring the circulating levels of NGF.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from severe burns

Exclusion Criteria:

* Major congenital malformations
* Antibiotic treatment 48 hours prior to admission
* Norepinephrine infusion > 0.5 mcg/k/min
* Lack of informed consent from parents or legal guardians

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from 1 month to 17 years of age suffering from severe burns, i.e. II/III degree and involving more than 8-10% of the body surface admitted to the Pediatric Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Qualitative description of NGF values in severely burned pediatric patients. | up to 30 days
  Patients will undergo blood sampling on days 2,7,14 and 30 after the traumatic event for the clinical follow-up envisaged by the internal protocol. A small aliquot of blood (5 ml) will be dedicated separately for the measurement of circulating NGF levels

SECONDARY OUTCOMES:
To evaluate the correlation of the extent of NGF expression with the severity of the burn and with the extent of the burned skin surface. | From date of inclusion in the study until 30 days after admission in pediatric intensive care
  In the protocol we will collect the following demographic and clinical variables: Age, gender, weight, total body surface area (%), Burn depth I II III degree, specific surface involvement (face, genitals, palms and soles), organ failure, use of inotropic and vasoconstrictor drugs, need for intubation and mechanical ventilation, quantification of fluid therapy for shock correction, infectious complications, need for surgery with possible homologous/autologous skin graft. these variables will be included to assess the correlation with NGF values

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio GC Conti, Professor, Principal Investigator — Fondazione Policlinico Gemelli IRCCS, Rome
Locations (1):
- Giorgio Conti, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We await the final analysis of the data to evaluate the definitive sharing of the collected data

REFERENCES:
- [Result] Pincelli C, Sevignani C, Manfredini R, Grande A, Fantini F, Bracci-Laudiero L, Aloe L, Ferrari S, Cossarizza A, Giannetti A. Expression and function of nerve growth factor and nerve growth factor receptor on cultured keratinocytes. J Invest Dermatol. 1994 Jul;103(1):13-8. doi: 10.1111/1523-1747.ep12388914. PMID 8027574
- [Result] Wu C, Boustany L, Liang H, Brennan TJ. Nerve growth factor expression after plantar incision in the rat. Anesthesiology. 2007 Jul;107(1):128-35. doi: 10.1097/01.anes.0000267512.08619.bd. PMID 17585224
- [Result] Matsuda H, Koyama H, Sato H, Sawada J, Itakura A, Tanaka A, Matsumoto M, Konno K, Ushio H, Matsuda K. Role of nerve growth factor in cutaneous wound healing: accelerating effects in normal and healing-impaired diabetic mice. J Exp Med. 1998 Feb 2;187(3):297-306. doi: 10.1084/jem.187.3.297. PMID 9449710
- [Result] Micera A, Vigneti E, Pickholtz D, Reich R, Pappo O, Bonini S, Maquart FX, Aloe L, Levi-Schaffer F. Nerve growth factor displays stimulatory effects on human skin and lung fibroblasts, demonstrating a direct role for this factor in tissue repair. Proc Natl Acad Sci U S A. 2001 May 22;98(11):6162-7. doi: 10.1073/pnas.101130898. Epub 2001 May 8. PMID 11344264